CLINICAL TRIAL: NCT05879549
Title: Comparison of Efficiency of Closed Kinetic Chain Exercises Versus Proprioceptive Exercises in Improving Balance and Gait in Patient With Hemophilia
Brief Title: Comparison of Efficiency of Closed Kinetic Chain Exercises Versus Proprioceptive Exercises Patient With Hemophilia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Tuğçe Poyraz İşleyen, Lecturer, Bahçeşehir University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-74555795-050.01.04-689576
Record Dates: First submitted 2023-05-05; First posted 2023-05-30 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: hemophilia; exercise; balance; proprioception
MeSH Terms: conditions — Hemophilia A; Hemophilia B; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Closed Chain Exercise Group (Experimental): Closed kinetic chain exercises will be given under the supervision of a physiotherapist, 2 sessions a week for 12 weeks.
  Interventions: Other: Closed Chain Exercise Group
- Proprioceptive Exercise Group (Experimental): Proprioceptive exercises will be given under the supervision of a physiotherapist, 2 sessions a week for 12 weeks.
  Interventions: Other: Proprioceptive Exercise Group
- Control Group (No Intervention): No intervention will be applied.

INTERVENTIONS:
Other: Closed Chain Exercise Group — Closed Chain Exercise Group
  Arms: Closed Chain Exercise Group
Other: Proprioceptive Exercise Group — Proprioceptive Exercise Group
  Arms: Proprioceptive Exercise Group

SUMMARY:
Hemophilia is a bleeding disorder caused by a deficiency of clotting factors in the blood. Muscle and joint bleeding are frequently observed in patients with hemophilia. Lower extremity bleeding can adversely affect balance, gait, and proprioception. The goal of this study; To compare the effectiveness of closed kinetic chain exercises and proprioceptive exercises on balance, proprioception and gait parameters in adolescent and young hemophilic individuals with lower extremity joint involvement.

The main question it aims to answer is:

Are the effects of closed kinetic chain exercises and proprioceptive exercises different on balance and walking in hemophilic individuals?

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with Hemophilia A and Hemophilia B
* Having a blood factor level below 5%,
* Between 13-25 years old
* History of bleeding to the lower extremity and target joint
* Total lower extremity Hemophilia joint health score ≥3
* Using prophylaxis

Exclusion Criteria:

* Having undergone lower extremity surgery in the last 6 months
* Having a Body Mass Index over 30 kg/m2
* Have an inhibitor
* Using a walking aid

Ages: 13 Years to 25 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 46 (Actual)
Dates: Start 2023-11-15 (Actual); Primary Completion 2024-03-30 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
Medio-lateral and Anterior-posterior stability index | 12 weeks
  Represents fluctuations from the horizontal around the mediolateral axis. Mediolateral sway and anterior-posterior stability will record in the double-leg stance for 20 seconds with Biodex Balance System. The feet are placed in a comfortable position for patients, and the center of gravity was recorded in the system to begin the test. Each test will repeat 3 times. A higher sway index indicates a decrease in postural stability.
walking speed | 12 weeks
  A 10-meter walking test will be used to evaluate walking.
Hemophilia joint health score | 12 weeks
  The HJHS is derived from a physical examination of the index joints by a health care professional who should have training and expertise in the conduct of a detailed musculoskeletal (MSK) examination. It is a measure of joint health and sits within the World . The current HJHS version 2.1 comprises an assessment of specific features, or items, of the six index joints and an assessment of global gait. For each of the six joints, the following items are scored: swelling (scored 0-3), duration of swelling (0-1), muscle atrophy (0-2), crepitus on motion (0-2), flexion loss (0-3), extension loss (0-3), joint pain (0-2), and strength (0-4). The maximum score for an individual index joint is 20. Gait is scored 0 to 4. The maximum HJHS total score is 124, with a higher score indicating worse joint health.

SECONDARY OUTCOMES:
Single leg stance test | 12 weeks
  The Single leg stance test (SLTS) measures static balance by challenging participants to stand unassisted on 1 leg. İndividuals stand for 30 or 45 seconds with their arms crossed across their chest or with their hands touching their hips. The SLST will completed with or without shoes and using the dominant or nondominant leg.
  The SLST will completed first with eyes open and then with eyes closed. Participants are timed as soon as their foot leaves the floor and stops once the foot touches the ground, the supporting foot shifts, their suspended foot touches the supporting leg, their eyes open in the eyes-closed trials, an arm is uncrossed or stops touching their hip, or if the maximum allotted time is reached.
  Three trials per condition are recorded, and either an average is calculated or the longest time is used. The SLST performance is reported in seconds (continuous) and requires a stopwatch.
Proprioception | 12 weeks
  A digital goniometer will be used to evaluate proprioception. The patient will be evaluated in a sitting position with eyes closed and open.
2-dimensional video-based gait kinematic analysis | 12 weeks
  2-dimensional video-based gait kinematic analysis is a simple, practical and inexpensive method in which a colour camera and passive markers are used. Firstly, the fifth metatarsophalangeal joint, the lateral malleolus, the lateral femoral condyle, and the trochanter major will marked as anatomical landmarks. Thereafter, passive markers will attached with double-sided adhesive tapes on the skin. Video recordswere then obtained with a high-speed 2D video camera. The camera will located on the tripod at a distance of 1.5 m from the patient, 0.86 m above the ground and with its optical axis perpendicular to the patients' sagittal axis. The patient will be asked to walk at a normal pace in front of the camera. The 2D records will processed using the Kinovea (version .8.15, Kinovea Open Source Project), which is a free 2D motion analysis will evaluate GKP. During the phases (midstance, preswing, midswing, and late swing phases) requiring a maximal ROMin the knee and ankle joints, kinematic

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tat NM, Tat AM, Oner AF, Karaman K, Kaplan S, Can F. Static postural balance evaluation and an investigation of the relationship with joint health in children with severe haemophilia: a controlled cross-sectional study. Haemophilia. 2021 Mar;27(2):e245-e252. doi: 10.1111/hae.14240. Epub 2021 Jan 24. PMID 33486846
- [Derived] Poyraz Isleyen T, Tarakci E, Leblebici G, Yeldan I, Zulfikar B. Comparison of Efficiency of Closed Kinetic Chain Exercises Versus Proprioceptive Exercises in Improving Balance and Gait in People With Hemophilia: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Apr 24;14:e66770. doi: 10.2196/66770. PMID 40273449